CLINICAL TRIAL: NCT01566123
Title: Clinical Phase I/II Trial to Investigate Preoperative Dose-Escalated Intensity-Modulated Radiation Therapy (IMRT) and Intraoperative Radiation Therapy (IORT) in Patients With Retroperitoneal Soft Tissue Sarcoma
Brief Title: Trial of Neoadjuvant Intensity-Modulated Radiation Therapy Followed by Surgery and Intraoperative Radiation Therapy in Resectable Retroperitoneal Soft Tissue Sarcoma (RETRO-WTS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RETROWTS
Record Dates: First submitted 2012-03-20; First posted 2012-03-29 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Retroperitoneal Soft Tissue Sarcoma
Keywords: retroperitoneal soft tissue sarcoma; IMRT; IORT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Neoadjuvant Intensity-Modulated Radiation Therapy Followed by Surgery and Intraoperative Radiation Therapy in Resectable Retroperitoneal Soft Tissue Sarcoma
  Interventions: Radiation: Neoadjuvant intensity-modulated radiation therapy (IMRT); Radiation: intraoperative radiation therapy (IORT)

INTERVENTIONS:
Radiation: Neoadjuvant intensity-modulated radiation therapy (IMRT) — neoadjuvant intensity-modulated radiation therapy, single dose 2.0-2.4 Gy, total dose 50-56 Gy
Radiation: intraoperative radiation therapy (IORT) — during surgery, 10-12 Gy (90% isodose) to the tumor bed or residual disease

SUMMARY:
Local control rates in patients with retroperitoneal soft tissue sarcoma (RSTS) remain disappointing even after gross total resection, mainly because wide margins are not achievable in the majority of patients. In contrast to extremity sarcoma, postoperative radiation therapy (RT) has shown limited efficacy due to its limitations in achievable dose and coverage. Although Intraoperative Radiation Therapy (IORT) has been introduced in some centers to overcome these dose limitations and resulted in improved outcome, local failure rates are still high even if considerable treatment related toxicity is accepted. As postoperative administration of RT has some general disadvantages, neoadjuvant approaches could offer benefits in terms of dose escalation, target coverage and reduction of toxicity, especially if highly conformal techniques like intensity-modulated radiation therapy (IMRT) are considered.

Therefore the RETROWTS trials has been designed as a prospective, one armed, single center phase I/II study investigating a combination of neoadjuvant dose-escalated IMRT (50-56 Gy) followed by surgery and IORT (10-12 Gy) in patients with at least marginally resectable RSTS. The primary objective is the local control rate after five years. Secondary endpoints are progression-free and overall survival, acute and late toxicity, surgical resectability and patterns of failure. The aim of accrual is 37 patients in the per-protocol population.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* histologically confirmed, primary or locally recurrent soft tissue sarcoma of the retroperitoneal space
* judged as at least marginally resectable
* absence of distant metastases
* tumor size ≥ 5 cm

Exclusion Criteria:

* missing written informed consent
* missing histological confirmation of soft tissue sarcoma
* Desmoid tumor (syn. aggressive fibromatosis)
* judged as gross incomplete or not resectable
* incomplete staging
* presence of distant metastases
* prior radiation therapy to the abdominal region
* participation in another clinical interventional study
* inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2007-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Local Control Rate | 5 year

SECONDARY OUTCOMES:
Progression free survival | up to 5 years from first day of treatment
Overall Survival | up to five years from first day of treatment
Acute toxicity | up to 3 months from first day of treatment
  scored according to CTCAE 3.0
Late Toxicity | up to 5 years after first day of treatment
  scored according to CTCAE 3.0 and RTOG criteria
Severe acute gastrointestinal toxicity | up to 3 months from first day of treatment
  severe defined as grade >= III, scored according to CTC AE 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, M.D., Ph.D., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Seidensaal K, Dostal M, Kudak A, Jaekel C, Meixner E, Liermann J, Weykamp F, Hoegen P, Mechtersheimer G, Willis F, Schneider M, Debus J. Preoperative Dose-Escalated Intensity-Modulated Radiotherapy (IMRT) and Intraoperative Radiation Therapy (IORT) in Patients with Retroperitoneal Soft-Tissue Sarcoma: Final Results of a Clinical Phase I/II Trial. Cancers (Basel). 2023 May 13;15(10):2747. doi: 10.3390/cancers15102747. PMID 37345084
- [Derived] Roeder F, Ulrich A, Habl G, Uhl M, Saleh-Ebrahimi L, Huber PE, Schulz-Ertner D, Nikoghosyan AV, Alldinger I, Krempien R, Mechtersheimer G, Hensley FW, Debus J, Bischof M. Clinical phase I/II trial to investigate preoperative dose-escalated intensity-modulated radiation therapy (IMRT) and intraoperative radiation therapy (IORT) in patients with retroperitoneal soft tissue sarcoma: interim analysis. BMC Cancer. 2014 Aug 27;14:617. doi: 10.1186/1471-2407-14-617. PMID 25163595
- [Derived] Roeder F, Schulz-Ertner D, Nikoghosyan AV, Huber PE, Edler L, Habl G, Krempien R, Oertel S, Saleh-Ebrahimi L, Hensley FW, Buechler MW, Debus J, Koch M, Weitz J, Bischof M. A clinical phase I/II trial to investigate preoperative dose-escalated intensity-modulated radiation therapy (IMRT) and intraoperative radiation therapy (IORT) in patients with retroperitoneal soft tissue sarcoma. BMC Cancer. 2012 Jul 12;12:287. doi: 10.1186/1471-2407-12-287. PMID 22788989